CLINICAL TRIAL: NCT04751578
Title: Abdominal Aortic Aneurysm Sac Healing and Prevention of Endoleaks - A Prospective Multicenter Study
Brief Title: Abdominal Aortic Aneurysm Sac Healing and Prevention of Endoleaks - Netherlands
Acronym: AAA-SHAPE_NLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shape Memory Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD1020
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: IMPEDE-FX Embolization Plug

INTERVENTIONS:
Device: IMPEDE-FX Embolization Plug — Fill an abdominal aortic aneurysm (AAA) sac outside of an endovascular aneurysm repair (EVAR) stent graft

SUMMARY:
To determine the safety and efficacy of IMPEDE-FX Embolization Plug and/or IMPEDE-FX Rapid Fill to fill an abdominal aortic aneurysm (AAA) sac outside of an endovascular aneurysm repair (EVAR) stent graft.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* A candidate for elective EVAR of an infrarenal aortic aneurysm ≥5.5 cm in diameter in men and ≥5.0 cm in women

Exclusion Criteria:

* An inability to provide informed consent
* Enrolled in another clinical study
* Aortoiliac aneurysm, or concomitant iliac artery ectasia or aneurysm (common iliac artery diameter >24 mm) close to the bifurcation and/or that cannot be adequately sealed
* Patent AAA sac feeding vessels (within the sac) >4 mm in diameter
* Volume of AAA sac to be filled after stent graft placement <20 mL or >135 mL, based on pre-procedure CTA (i.e. aortic flow volume exclusive of stent graft volume)
* Use of aortic stent grafts other than the Gore Excluder AAA Endoprosthesis, Cook Zenith Flex AAA Endovascular Graft, or Medtronic Endurant II Stent Graft to treat the AAA
* Planned use of the chosen stent graft outside its instructions for use (IFU)
* Planned use of fenestrated or chimney stent grafts
* Study participants in which stent graft placement is abandoned for any reason, and/or in which the investigator decides, during the course of the stent graft placement, that the study procedure may not be appropriate
* Planned use of embolic devices other than the investigational product to embolize the AAA sac
* Vascular disease and/or anatomy that preclude the safe access and positioning of a catheter to deliver the investigational product into the AAA sac
* Ruptured, leaking, or mycotic (infected) aneurysm
* Aneurysmal disease of the descending thoracic aorta
* Coagulopathy or uncontrolled bleeding disorder
* Long-term (>6 months prior to the procedure) use of direct oral anticoagulant or any vitamin K antagonist anticoagulant use
* Serum creatinine level >2.5 mg/dL;
* Cerebrovascular accident within 3 months prior to the procedure
* Myocardial infarction and/or major heart surgery within 3 months prior to the procedure
* Atrial fibrillation that is not well rate controlled
* Unable or unwilling to comply with study follow-up requirements
* Life expectancy of <2 years post-procedure
* Known hypersensitivity or contraindication to platinum, iridium, or polyurethane
* A condition that inhibits radiographic visualization during the implantation procedure
* History of allergy to contrast medium that cannot be managed medically
* Uncontrolled co-morbid medical condition, including mental health issues, that would adversely affect participation in the study
* Pregnant or a lactating female. For females of child-bearing potential, based on a positive pregnancy test within 7 days prior to the procedure or refusal to use a medically accepted method of birth control for the duration of the study
* Prisoner or member of other vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of related major adverse events (MAEs) | 30 days post-procedure
  Incidence of related major adverse events (MAEs)
Efficacy - Technical Success | Immediately after the intervention
  Technical success, defined as filling of the residual flow lumen of the AAA sac with investigational products

SECONDARY OUTCOMES:
Incidence of related major adverse events (MAEs) | 5 years post-procedure
  Incidence of related major adverse events (MAEs)
Incidence of related serious adverse events (SAEs) | 5 years post-procedure
  Incidence of related serious adverse events (SAEs)
Efficacy - Type II endoleaks | 5 years post-procedure
  Incidence of type II endoleaks
Efficacy - Type I and type III endoleaks | 5 years post-procedure
  Incidence of type I and type III endoleaks
Efficacy - AAA sac diameter/volume | 5 years post-procedure
  Change in AAA sac diameter/volume
Efficacy - Open repair | 5 years post-procedure
  Rate of conversion to open AAA repair
Efficacy - Reinterventions | 5 years post-procedure
  Rate of other reinterventions related to the AAA sac growth and/or complications

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - ETZ Elisabeth, Tilburg, Tilburg

IPD SHARING:
Plan to Share IPD: No